CLINICAL TRIAL: NCT05896137
Title: A Phase II Study to Evaluate Safety, Tolerability and Efficacy, of CS0159 in Patients Subjects With Primary Sclerosing Cholangitis, Multicenter, Randomized, 12-week Double-blind, Placebo-controlled, and 40-week Open Study
Brief Title: CS0159 in Chinese Patients With PSC (Primary Sclerosing Cholangitis)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSC-CS0159-003
Record Dates: First submitted 2023-05-18; First posted 2023-06-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2mg CS0159 (Experimental): CS0159 tablet 2mg for 12 weeks
  Interventions: Drug: CS0159
- 4mg CS0159 (Experimental): CS0159 tablet 4mg for 12 weeks
  Interventions: Drug: CS0159
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Drug: CS0159

INTERVENTIONS:
Drug: CS0159 — Oral QD
  Other Names: Pleacbo

SUMMARY:
A phase II Study of CS0159 in Chinese patients with PSC(Primary Sclerosing Cholangitis)

DETAILED DESCRIPTION:
A phase II study to evaluate safety, tolerability and efficacy, of CS0159 in patients with Primary Sclerosing Cholangitis, this is a multicenter, randomized, 12-weeks double-blind, placebo-controlled, and 40-week open study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age≥18 or age≤75 years when sign ICF
2. Within the last year, have a clinical diagnosis of PSC with a consistent magnetic resonance cholangiopancreatography (MRCP) orendoscopic retrograde cholangiopancreatography (ERCP) Prcutaneous Transhepatic Cholangiography(PTC) showing sclerosing cholangitis
3. 1.50×ULN≤ALP≤10×ULN, and TBil≤3×ULN during screen
4. Taken UDCA(≤25mg/kg/d)≥6 months before randomization and stable does≥ 3 months, or not used UDCA≥3 months before randomization
5. For subject with a history of IBD

   1. Patients with Crohn's Disease (CD),Must be in remission, CDAI<150 or CDAI of score ≤4
   2. Patients with(Ulcerative Colitis)UC,Must be in remission or only mild activity,Some Mayo scores range from 0 to 4
6. Be able to understand and Comply with the study protocol sign a written informed consent form(ICF)voluntarily

Exclusion Criteria,

1. Presence of documented secondary sclerosing cholangitis when screening,or direct evidence IgG4 related sclerosing cholangitis or serum IgG4 ≥ 4 ×ULN
2. Small duct PSC
3. ALT or AST>5×ULN
4. Taken( ObeticholicAcid) OCA within 3 months before randomization
5. Acute cholangitis was suspected or confirmed within 3 months prior to randomization, Including acute cholangitis being treated during screening
6. Presence of percutaneous drain or bile duct stent at the time of screening or during the study
7. Known concurrent comorbidities with other hepatobiliary diseases including, but not limited to: active hepatitis B virus or hepatitis C virus infection (see Exclusion Criterion 9), primary biliary cholangitis, complete biliary obstruction, acute cholecystitis or gallstones with significant symptoms, Autoimmune Hepatitis (AIH) or overlap with other autoimmune liver diseases, Alcoholic Hepatitis, Non-Alcoholic Steatohepatitis, Suspected or Diagnosed Primary Hepatocellular Cancer, and Bile Duct Cancer;
8. Child-Pugh patients with grade B or C cirrhosis,Present complications related to cirrhosis or End-stage liver disease ,Including history of liver transplantation Preparing for liver transplantation (Model for End-Stage Liver Disease)MELD≥15，Portal hypertension complications,Complications of cirrhosis
9. Patients who are HBsAg-positive, HCVAb-positive, HIVAb-positive or TPAb-positive at screening
10. Cr(Creatinine)≥1.5×ULN also Cr(Creatinine)clearance rate<60 mL/min
11. PLT(Platelet)<80×10^9/L
12. INR(international normalized ratio)>1.3
13. ALB<3.5g/dL
14. Severe pruritus may require systemic medication Within 2 months prior to randomization
15. Arrhythmia,male QTc≥450 ms,female QTc≥470 ms, during screening
16. A disease that interferes with the absorption, distribution, metabolism, or excretion of a test drug,such as moderate to severe activity IBD patient, Previous gastric bypass surgery
17. Moderate or intense inhibition of CYP3A4 was performed during 14 days prior to randomization and throughout the trial Preparation or inducer
18. The presence of diseases that may cause non-hepatic elevation of ALP (e.g. Paget's disease) or may cause it Diseases with a life expectancy of less than 2 years
19. History of malignancy within the past 5 years prior to randomization
20. Immunosuppressants, budesonide, and other systemic glucocorticoids were used within 28 days before randomization and throughout the clinical study period;
21. Use of fenofibrate or another fibrate within 28 days prior to randomization and throughout the clinical study period; Hepatotoxic drugs; Hepatoprotective drugs and other hepatoprotective drugs were given stable doses <28 days before randomization or could not maintain stable doses during the trial; cholagogue
22. Interleukin or other cytokines were used 12 months before randomization and throughout the trial Or antibodies to chemokines or immunotherapy
23. Drug and/or alcohol abuse within the first six months of randomization
24. Poor blood pressure control,systolic pressure>160 mmHg or dpb >100 mmHg
25. Poor blood sugar control,Glycated hemoglobin>9.0%
26. Females who are pregnant or plan to pregnant,Fertile but refusing to sign informed consent, or breastfeed
27. Participated any other study within 30 days prior randomization,and received other experimental medications therapy
28. It is unsuitable to participate for the study or has other diseases by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
AE incidence | Baseline to 12 weeks
  AE incidence in placebo, 2mg and 4mg group
relative changes from baseline in ALP at week 12 | Baseline to 12 weeks
  The reduction of percentage of ALP level from baseline to 12 weeks

SECONDARY OUTCOMES:
Absulute changes from baseline in ALP at week 12 | Baseline to 12 weeks
  The reduction of ALP level from baseline to 12 weeks
ALP and TBil changes | Baseline to 12 weeks
  Compared with placebo, ALP< 1.50 ULN, (total bilirubin) TBil ≤ULN
TBA changes | from basline to 12 weeks, and to 40 weeks
  BA change from baseline
Pruritus incidence | from basline to 40 weeks
  changes from baseline in the study period

CONTACTS AND LOCATIONS:
Overall Officials: Rong Deng, Study Director — Cascade Pharmaceuticals, Inc
Locations (11):
- China (11):
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Friendship Hospital, Captail Medcial University, Beijing, Beijing Municipality
  - Beijing YouAn Hostital, Captial Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - The Seconed Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shaoyifu Hospital of Zhejiang University Medical, Hangzhou, Zhejiang
  - The First Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No